CLINICAL TRIAL: NCT05480943
Title: Prevalence of Thiamine Deficiency in Hospitalized Non-Alcoholic Veterans
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Sierra Nevada Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: F4101-P; IRBNet ID 1867369-3 (Other: VA Sierra Nevada Health Care System)
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Thiamine Deficiency; Thiamine Deficiency; Sequelae
Keywords: thiamine deficiency; Wernicke's encephalopathy; beriberi; delirium; polyneuropathy; vitamin B1; falls
MeSH Terms: conditions — Thiamine Deficiency; Wernicke Encephalopathy; Beriberi; Delirium; Polyneuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — No specimen will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized non-alcoholic Veterans: Any Veteran with full admission to the VA Sierra Nevada Healthcare System Hospital.
  Interventions: Dietary Supplement: Thiamine repletion

INTERVENTIONS:
Dietary Supplement: Thiamine repletion — If a participant is determined by clinical characteristics or biomarker results to be thiamine deficient, thiamine supplementation was provided.

SUMMARY:
Thiamine micronutrient deficiency (TD) can cause a variety of non-specific symptoms and leads to several thiamine deficiency disorders such as heart failure, polyneuropathy, Wernicke's Encephalopathy and generalized weakness and debility. Symptoms are often vague and non-specific such as fatigue, leg swelling, imbalance, confusion, mood disorders, gastrointestinal upset, and weakness. Hospitalized Veterans may be particularly susceptible to TD due to food insecurity and chronic illnesses which cause inflammation and increased metabolic demands. This study aims to determine the prevalence of TD in hospitalized Veterans which has never been done before. The investigators also seek to identify risk factors causing TD including acute and chronic forms of inflammation, food insecurity, and dietary habits. Lastly, the investigators hope to clarify the abnormally low levels of blood thiamine that correlate with symptoms of TD that improve with replenishment.

DETAILED DESCRIPTION:
Background: Thiamine deficiency (TD) causes a variety of thiamine deficiency disorders (TDDs) such as neuropsychiatric disturbances, polyneuropathy, ataxia, weakness and falling, and non-ischemic heart failure. Left untreated, TD can be associated with poor quality of life, loss of independence, and inability to complete activities of daily living. The prevalence of TD in non-alcohol using hospitalized Veterans is not known but is probably much higher than the general population. Loss of functional ability leads to increased need for rehabilitation.

The objective of this proposal is to measure the prevalence of TDDs in Veterans who do not use excess alcohol who are ill enough to require hospitalization, determine if inflammation increases the risk of developing TD, and determine the optimal cutoff points for two biomarkers of TD to diagnose of TDDs. The central hypothesis is that TD prevalence is as high as 25% in hospitalized non-alcoholic Veterans, far greater than the historically reported prevalence of 3% or less, and that TDD's occur in the "low normal" range of current cutoff values for available thiamine bioassays. A secondary hypothesis is that inflammatory conditions, which are known to cause cachexia and malnutrition, put hospitalized Veterans at increased risk as they often present with acute inflammatory conditions. The rationale underlying this proposal is that hospital practitioners currently underdiagnose and undertreat TDDs which leads to continued morbidity and loss of function. If the hypothesis is correct that the prevalence is as high as 25%, this knowledge will increase awareness of the problem and lead practitioners to diagnose and treat them more often. In addition, clarifying the "abnormally low" biomarker cutoff levels by measuring them in Veterans with TDDs is very important as the current "normal" ranges were determined in healthy volunteers. The central hypothesis will be tested by pursuing three specific aims: 1) determine the prevalence of TD, as defined by whole blood and plasma thiamine levels together with symptom responsive disease in consecutively hospitalized medicine patients who do not use excessive alcohol; 2) define TDDs as cases with low or "low normal" thiamine levels and symptoms that improve with thiamine replenishment; 3) determine if acute and chronic inflammatory conditions with elevated biomarkers of inflammation increase the risk of developing TDD. The investigators expect to find the prevalence of TD is closer to 25% and that the low end of "normal" biomarker levels as published by reference laboratories is too low, missing a percentage of TDDs.

Research design: To accomplish these aims, the investigators will utilize a prospective cohort study design to determine the prevalence of TD in consecutively hospitalized non-alcoholic medicine patients, as defined by low or "low normal" thiamine biomarker levels and thiamine responsive symptoms. Nested within this the investigators will conduct an open label treatment study with those exhibiting symptoms and define TDDs as cases with low or "low normal" thiamine levels and symptoms of TD that improve with thiamine administration. Lastly, utilizing a nested case control study design with cases being those with a TDD and controls being asymptomatic Veterans with normal biomarkers, determine if acute and chronic inflammatory conditions with elevated biomarkers of inflammation increase the risk of developing TDDs.

ELIGIBILITY:
Inclusion Criteria:

* full admission to the hospital medical service (not on observation status)

Exclusion Criteria:

* excess alcohol intake as defined by the National Institute of Alcohol Abuse and Alcoholism
* taking thiamine supplement
* quadriplegic
* lives more than 75 miles from the medical center
* unable to demonstrate capacity to understand the study and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who are admitted to the medicine service at the VA Sierra Nevada Healthcare System hospital in Reno, NV who do not use alcohol to excess. The Veterans will need to live within 75 miles of the medical center to facilitate return for follow up appointments.
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth A Mates, MD PhD, Principal Investigator — VA Sierra Nevada Health Care System, Reno, NV
Locations (1):
- VA Sierra Nevada Health Care System, Reno, NV, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data set will be shared upon request made to Dr. Elisabeth Mates

REFERENCES:
- [Background] Mates E, Alluri D, Artis T, Riddle MS. A Retrospective Case Series of Thiamine Deficiency in Non-Alcoholic Hospitalized Veterans: An Important Cause of Delirium and Falling? J Clin Med. 2021 Apr 1;10(7):1449. doi: 10.3390/jcm10071449. PMID 33916273
- [Background] Gomes F, Bergeron G, Bourassa MW, Fischer PR. Thiamine deficiency unrelated to alcohol consumption in high-income countries: a literature review. Ann N Y Acad Sci. 2021 Aug;1498(1):46-56. doi: 10.1111/nyas.14569. Epub 2021 Feb 11. PMID 33576090
- [Background] Donnino MW, Carney E, Cocchi MN, Barbash I, Chase M, Joyce N, Chou PP, Ngo L. Thiamine deficiency in critically ill patients with sepsis. J Crit Care. 2010 Dec;25(4):576-81. doi: 10.1016/j.jcrc.2010.03.003. Epub 2010 Jun 19. PMID 20646908
- [Background] Whitfield KC, Bourassa MW, Adamolekun B, Bergeron G, Bettendorff L, Brown KH, Cox L, Fattal-Valevski A, Fischer PR, Frank EL, Hiffler L, Hlaing LM, Jefferds ME, Kapner H, Kounnavong S, Mousavi MPS, Roth DE, Tsaloglou MN, Wieringa F, Combs GF Jr. Thiamine deficiency disorders: diagnosis, prevalence, and a roadmap for global control programs. Ann N Y Acad Sci. 2018 Oct;1430(1):3-43. doi: 10.1111/nyas.13919. Epub 2018 Aug 27. PMID 30151974
- [Background] Lee DC, Chu J, Satz W, Silbergleit R. Low plasma thiamine levels in elder patients admitted through the emergency department. Acad Emerg Med. 2000 Oct;7(10):1156-9. doi: 10.1111/j.1553-2712.2000.tb01268.x. PMID 11015250
- [Background] Smith TJ, Johnson CR, Koshy R, Hess SY, Qureshi UA, Mynak ML, Fischer PR. Thiamine deficiency disorders: a clinical perspective. Ann N Y Acad Sci. 2021 Aug;1498(1):9-28. doi: 10.1111/nyas.14536. Epub 2020 Dec 10. PMID 33305487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All admissions to the hospital were screened and Veterans were excluded if they reported excess alcohol intake; taking thiamine; lived more than 70 miles from the hospital. Those who passed screening were approached for consent. If they were unable to comprehend and "read back" basic elements of the informed consent (as determined by the U-ARE protocol), they were not included due to prohibitive state laws. The first patient was enrolled on July 19, 2022. The last Veteran was enrolled 8/27/2024.
Pre-assignment Details: 1713 participants were screened. Of those, 336 were being discharged too soon for study procedures, 322 lived too far away, 211 took thiamine, 149 had alcohol use disorder, 134 were excluded for reasons due to study logistics (e.g. lack of provider to complete exams, patient too busy, etc.), and 99 cognitively could not consent. Of the remaining, 256 did not want to participate and 206 were enrolled.
Groups:
- Veterans Without Alcohol Use Disorder Admitted to the Hospital: Veterans with full admission to the hospital who did not have alcohol use disorder, lived within 70 miles of the hospital, were able to read back key portions of the consent, and who were not taking thiamine supplements.
Period: Evaluation for Thiamine Deficiency
Arm/Group | Veterans Without Alcohol Use Disorder Admitted to the Hospital
Started | 206
Obtained Plasma Thiamine Results | 181 (12 were either discharged before phlebotomy or had invalid lab results, 7 were subsequently found to take a B-complex or thiamine supplement, 3 were given thiamine by their inpatient provider before phlebotomy, one was subsequently found to drink excess alcohol, one revoked consent before phlebotomy, and one was given a large volume blood transfusion which can alter thiamine levels. That left 181 participants remaining the in the study.)
Answered Interview Questions (4 did not complete interviews due to refusal, discharge before completion, or too busy with procedures to complete of which 1 completed physical exam) | 177
Completed Initial Physical Exam (19 missed physical exam either due to refusal or discharge prior to procedure completed) | 162
Completed | 162
Not Completed | 44
Not completed — Lost to Follow-up | 31
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 1
Period: Suspected Thiamine Deficiency
Arm/Group | Veterans Without Alcohol Use Disorder Admitted to the Hospital
Started | 124 (124 of the 162 that completed physical exams had clinical or biomarker evidence of thiamine deficiency and were prescribed thiamine repletion and invited back for reevaluation.)
Completed | 60
Not Completed | 64
Not completed — Lost to Follow-up | 64

BASELINE CHARACTERISTICS:
Groups:
- Hospitalized Non-alcoholic Veterans: Veterans with full admission to the VA Sierra Nevada Healthcare System Hospital who do not have alcohol use disorder (AUD).
Arm/Group | Hospitalized Non-alcoholic Veterans
Number analyzed (Participants) | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.33 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 193
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 175
  More than one race | 1
  Unknown or Not Reported | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 206
Plasma thiamine level [Count of Participants; unit: Participants] — Plasma thiamine level less than 8 nmol/L were considered low Population: 181 with plasma thiamine biomarker results
  Participants
    Low plasma thiamine: number analyzed (Participants) | 181
    Low plasma thiamine | 49
    Normal plasma thiamine: number analyzed (Participants) | 181
    Normal plasma thiamine | 132
Highly sensitive C-reactive protein [Count of Participants; unit: Participants] — Participants with highly sensitive C-reactive protein levels greater than 1.0 mg/dL were considered abnormal / elevated consistent with inflammation. Population: Only 125 participants had C-reactive protein lab results
  Participants
    Normal C-reactive protein: number analyzed (Participants) | 125
    Normal C-reactive protein | 38
    Elevated C-reactive protein: number analyzed (Participants) | 125
    Elevated C-reactive protein | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Thiamine Deficiency (Low Plasma Thiamine) Out of Total Number of Enrolled Veterans With Plasma Thiamine Results
Description: The percentage of enrolled non-alcoholic veterans who have thiamine deficiency (defined as low plasma thiamine levels) out of the total number of enrolled Veterans with plasma thiamine results.
Time Frame: Baseline
Population: Enrollees with plasma thiamine levels
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Veterans With Plasma Thiamine Results: Enrolled Hospitalized non-alcoholic Veterans with plasma thiamine results.
Arm/Group | Enrolled Veterans With Plasma Thiamine Results
Number analyzed (Participants) | 181
Participants | 49

2. Secondary Outcome: Association of Thiamine Deficiency and Inflammation
Description: Determine if there is an association between thiamine deficiency defined by low plasma thiamine levels, and elevated highly sensitive C-reactive protein indicating inflammation.
Time Frame: Baseline
Population: Participants with results of both plasma thiamine level and C-reactive protein who were thiamine deficient were analyzed to determine if there was an association between thiamine deficiency and increased inflammation.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Veterans With Both Plasma Thiamine and CRP Results Who Were Thiamine Deficient: Veterans with both thiamine biomarker and highly sensitive C-reactive protein biomarker results who were thiamine deficient.
Arm/Group | Enrolled Veterans With Both Plasma Thiamine and CRP Results Who Were Thiamine Deficient
Number analyzed (Participants) | 33
Participants
  Normal CRP | 8
  Elevated CRP | 25
Statistical Analysis 1: Comparison: Enrolled Veterans With Both Plasma Thiamine and CRP Results Who Were Thiamine Deficient; For the subset of 123 participants with both C-reactive protein level and plasma thiamine levels (125 had C-reactive protein results but 2 were missing plasma thiamine levels), we used Chi-Square to test for association between those who were thiamine deficient and had elevated C-reactive protein (CRP) levels. A priori hypothesis was that inflammation would cause thiamine deficiency due to increased metabolic demands; Test type: Other — chi-square tested correlation between CRP and thiamine deficiency; p = 0.6097, Chi-squared — P<=0.05 considered significant

3. Secondary Outcome: Cut-point Analysis of Thiamine Biomarkers
Description: The investigators will determine the low end of normal thiamine levels in veterans with treatment-responsive thiamine deficiency symptoms using a composite score to compare exam findings before and after treatment with thiamine.
Time Frame: Baseline compared to follow up visit
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: two months
Groups:
- Hospitalized Non-alcoholic Veterans: Veterans with full admission to the hospital who did not have alcohol use disorder, lived within 70 miles of the hospital, were able to read back key portions of the consent, and who were not taking thiamine supplements.
Arm/Group | Hospitalized Non-alcoholic Veterans
All-Cause Mortality (participants affected / at risk) | 23/181
Serious Adverse Events (participants affected / at risk) | 0/181
Other Adverse Events (participants affected / at risk) | 1/181
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hospitalized Non-alcoholic Veterans (N=181)
Diarrhea (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Multiple prolonged work stoppages due to unforeseen events led to lower than expected enrollment. Poor compliance with follow up visits after initial evaluation in the hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT05480943/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05480943/ICF_000.pdf